CLINICAL TRIAL: NCT06178029
Title: Effectiveness of Acupuncture Treatment Applied in Addition to the Rehabilitation Program in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Zeynep İnce, Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10026391
Record Dates: First submitted 2023-11-06; First posted 2023-12-20 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: Acupuncture; Gait; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional rehabilitation (Active Comparator): 20 multiple sclerosis patients will receive conventional rehabilitation
  Interventions: Other: Conventional Rehabilitation
- conventional rehabilitation and acupuncture (Active Comparator): 20 multiple sclerosis patients will receive conventional rehabilitation and acupuncture treatment.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — 20 patients with multiple sclerosis meeting the criteria will undergo conventional rehabilitation and acupuncture treatment.
  Arms: conventional rehabilitation and acupuncture
Other: Conventional Rehabilitation — 20 patients with multiple sclerosis meeting the criteria will undergo conventional rehabilitation
  Arms: conventional rehabilitation

SUMMARY:
The purpose of the study is to assess the effect of acupuncture treatment combinated with conventional rehabilitation methods on gait, fatigue, quality of life and bladder functions in patients with multiple sclerosis

DETAILED DESCRIPTION:
After being informed about study and potential risks, all patient giving written informed consent will undergo screening period determine eligibility for study entry. The patients who meet the eligibility recruitments will get treatment into two groups in a conventional rehabilitation and acupuncture combined with conventional rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MS according to McDonald criteria
* EDSS score between 1-6
* The patient is clinically stable
* Having not had a new MS attack in the last 3 months
* Being cognitively suitable to participate in the study

Exclusion Criteria:

* Being clinically unstable
* Inability to cognitively participate in tests
* Having received acupuncture treatment in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Timed 25 Foot Walk Test Score | Baseline, after 1 month and 3 month changes
  The Timed 25 Foot Walk test assesses a patient's ability to walk 25 feet distance.Patient's walking speed in m/s calculate

SECONDARY OUTCOMES:
Neurogenic Bladder Symptom Scoring | Baseline, after 1 month and 3 month changes
  The Neurogenic Bladder Symptom Score (NBSS) is a validated 24 item questionnaire that measures bladder symptoms across 3 different domains: incontinence (scored 0-29), storage and voiding (scored 0-22), and consequences (scored 0-23); there is a single general urinary QOL question scored from 0 (pleased) to 4 (unhappy). For all domains, a higher score represents a worse symptom burden or QOL
Incontinence Quality of Life Questionnaire | Baseline, after 1 month and 3 month changes
  There are 22 questions. The 22 items can be further grouped into 3 subscales: Avoidance and Limiting Behaviour (8 items), Psychosocial Impacts (9 items), and Social Embarrassment (5 items). The total I-QOL and 3 subscale scores are calculated by summing the unweighted item score and transforming them to a 100 point scale where 0 = most severe, and 100 = no problem . The instrument has been widely used and has been successfully validated for people with uriner incontinence
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Baseline, after 1 month and 3 month changes
  The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument
Fatigue Severity Scale | Baseline, after 1 month and 3 month changes
  The FAS is a 10-item scale evaluating symptoms of chronic fatigue. As the score increases in FAS, the severity of the patient's fatigue also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep İNCE KESKİN, Medical Doctor, Principal Investigator — Ankara City Hospital Bilkent; Müyesser ARAS, Professor Doctor, Study Director — Ankara City Hospital Bilkent; Semra MUNGAN, Associate Professor, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Bilkent-Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Criado MB, Santos MJ, Machado J, Goncalves AM, Greten HJ. Effects of Acupuncture on Gait of Patients with Multiple Sclerosis. J Altern Complement Med. 2017 Nov;23(11):852-857. doi: 10.1089/acm.2016.0355. Epub 2017 Apr 14. PMID 28410453